CLINICAL TRIAL: NCT06912841
Title: Deep Brain Stimulation (DBS) MatchMaker
Acronym: DBSMatchMaker
Status: Enrolling by invitation | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Darius Ebrahimi-Fakhari, Darius Ebrahimi-Fakhari, MD, PhD, Boston Children's Hospital
Other Study IDs: IRB-A00047069
Record Dates: First submitted 2024-12-27; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: TOR1A; PANK2; HPRT1; EIF2AK2; SOX2; KMT2B; GABRB2; ADCY5; UBA5; GNAO1; SGCE; TNPO2; GNB1; PLA2G6; Movement Disorders; Dystonia; Chorea
Keywords: Deep Brain Stimulation; DBS; movement disorders; dystonia; genetic
MeSH Terms: conditions — Movement Disorders; Dystonia; Chorea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
DBS Matchmaker (https://www.dbsmatchmaker.com) is a platform designed to connect clinicians worldwide who are treating rare movement disorders with deep brain stimulation (DBS). It facilitates global collaboration and knowledge sharing to enhance patient care by improving patient selection, counseling, treatment, and outcomes for individuals with movement disorders.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) is an effective treatment for childhood-onset dystonia and other hyperkinetic disorders, with emerging evidence supporting its use in an expanding range of monogenic movement disorders. While some conditions, such as TOR1A-related dystonia, are well-established indications for DBS, many rare and ultra-rare movement disorders are also being considered for treatment. However, individual centers often have limited experience with these conditions, leading to mostly anecdotal observations. Furthermore, the published literature is often scarce or not up to date.

To bridge this gap, DBSMatchMaker (https://www.dbsmatchmaker.com) was developed both as a tool to assist clinicians in determining the appropriateness of DBS for their patients, and in supporting therapy adjustments for patients who already have an implant. By connecting specialists worldwide, DBSMatchMaker seeks to improve patient selection, counseling, treatment, and outcomes for individuals with rare movement disorders, ultimately enhancing care for this underserved patient population.

By connecting specialists worldwide, the platform aims to:

Improve patient selection and counseling; Enhance treatment strategies and outcomes for individuals with rare movement disorders; Ultimately, DBSMatchmaker seeks to elevate the standard of care for this underserved patient population.

Key Features:

Global Collaboration: Enables clinicians to connect with peers treating similar conditions with DBS, fostering a worldwide network of specialists.

Knowledge Sharing: Facilitates the exchange of experiences and expertise in DBS treatment, promoting collaborative learning.

Enhanced Patient Care: Aims to improve treatment outcomes through shared insights and collective knowledge.

How It Works:

Clinicians can submit information about their cases to DBS Matchmaker. The platform adheres to strict safety and privacy protocols; it does not collect identifiable data, and the database is not searchable by users. Submitted data may be shared with potential collaborators to facilitate connections between medical centers treating similar cases.

Developed by the Ebrahimi-Fakhari Laboratory at Boston Children's Hospital, DBS Matchmaker is committed to advancing the care of individuals treated with DBS for rare movement disorders.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of all ages with genetic movement disorders, who are undergoing or being considered for DBS treatment.

Exclusion Criteria:

* Individuals who have not undergone DBS treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of individuals with rare genetic movement disorders characterized by childhood-onset dystonia and other hyperkinetic disorders. Cases involve individuals being considered for or undergoing treatment with deep brain stimulation (DBS).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Identify Potential Matches | 5 years
  Clinicians can submit their DBS cases through a secure platform (https://www.dbsmatchmaker.com/), which are then reviewed to identify potential matches with other centers treating similar cases. When a match is found, direct connections between medical teams are facilitated to promote collaboration and knowledge sharing.
Connect Clinicians & Facilitate Collaboration | 5 years
  DBS Matchmaker is a platform designed to connect clinicians worldwide who are treating rare movement disorders with deep brain stimulation (DBS). It facilitates global collaboration and knowledge sharing to enhance patient care.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.dbsmatchmaker.com/